CLINICAL TRIAL: NCT04160754
Title: Mindfulness for at Risk Youth: Understanding Substance Use and Important Mechanisms of Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jordan Davis, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: up-18-00230
Record Dates: First submitted 2018-10-03; First posted 2019-11-13 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Use, Underage; Alcohol Problem Drinking; Substance Use
Keywords: Trauma; Delinquency; Substance Use; Emotion Regulation; Impulsivity; Executive Functioning
MeSH Terms: conditions — Underage Drinking; Alcoholism; Substance-Related Disorders; Wounds and Injuries; Emotional Regulation; Impulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBRP (Experimental): The experimental group will receive treatment as usual plus eight Mindfulness based relapse prevention (MBRP) therapy sessions.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention
- Control (CTL) (Active Comparator): The CTL group will receive treatment as usual plus information on the neurobiology of addiction and healthy behaviors.
  Interventions: Behavioral: Control (CTL)

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention — Individuals assigned to the experimental group will receive interventions normally provided at the clinic and eight 1.5-hour group sessions of MBRP. Each sessions will occur once per week and will target a specific theme such as being aware of personal triggers, maintaining present focus, allowing or letting things be, responding to emotional and physical experiences in skillful ways, and recognizing intrusive thoughts. Each session will incorporate a mindfulness meditation technique (e.g.,SOBER breathing space and "urge surfing"). Participants will receive materials (e.g., recordings) with which to perform practices and meditation during the intervention phase.
  Arms: MBRP
Behavioral: Control (CTL) — Individuals assigned to the CTL group will receive interventions provided at the clinic and up to eight CTL sessions. The CTL group will receive information (reading) and videos once per week on health behaviors (e.g., exercise, eating) and the neurobiology of addiction. This approach will reduce the possibility that intervention effects are solely due to the experimental group's receiving extra attention. In contrast to the active intervention, sessions will be educational in nature, with no motivational, cognitive, or behavioral components
  Arms: Control (CTL)

SUMMARY:
This study will be the first to explore mindfulness as a prevention intervention among transition age youth and those with previous involvement in the juvenile or criminal justice system with substance use problems and history of exposure to violence/trauma. The study will focus on preventing escalation of substance use (e.g., alcohol and marijuana), trauma symptoms, and recidivism by using an intervention to target self-regulation and executive functioning.

Justice involved youth have higher rates of alcohol use and related consequences and higher rates of exposure to violence (Post Traumatic Stress Disorder) compared to their non-justice involved peers. Prior research has found aspects of self-regulation (emotion regulation, impulse control), stress, and craving to be important putative targets in reducing alcohol use. With high rates of recidivism and increased risk of long term problems associated with substance use, it is imperative to test interventions that can reach at risk youth and target both alcohol use and important psychological and neurocognitive self-regulation mechanisms.

This study tests whether the use of Mindfulness-Based Relapse Prevention (MBRP) for at risk young adults results in changes in important self-regulation mechanisms and improved alcohol use outcomes. Individuals assigned to the experimental group will receive interventions normally provided at a community clinic and eight 1.5-hour group sessions of MBRP. Sessions will occur once per week. Each session will target a specific theme such as being aware of personal triggers, maintaining present focus, allowing or letting things be, responding to emotional and physical experiences in skillful ways, and recognizing intrusive thoughts. Further, each session will incorporate a mindfulness meditation technique.

The central hypothesis will be tested through a focus on three specific aims: (1) Beta pilot testing and refining MBRP based on feedback from focus groups, (2) testing the efficacy of MBRP on substance use outcomes compared to an active control, and (3) assessing mechanisms of change for MBRP including self-regulation and neurocognitive facets such as working memory and inhibition.

DETAILED DESCRIPTION:
The long-term goal of this proposal is to improve alcohol use outcomes by targeting emotion regulation (ER), impulsivity (IMP), and executive functioning (EF) constructs among racially and ethnically diverse (primarily Hispanic and Black) at risk young adults. With a similar population, the investigators pilot tested a novel Mindfulness-Based Intervention (MBI), Mindfulness-Based Substance Abuse Treatment for Adolescents (MBRP) with with marginalized young adults. Findings from adolescent samples have found support for the intervention's effect on problem behaviors, decision making, and self-esteem. However, extent research in this area has not assessed substance use or self-regulation. In a sample of marginalized young adults receiving treatment at a residential treatment facility, MBRP was found to significantly decrease stress and substance use outcomes. In addition, only one study has investigated the effect of a MBI on neurocognitive functioning with justice-involved youth. Unfortunately, this was not a clinical intervention and did not assess EF as a mechanism of change. The current study proposes to recruit 70-80 young adults (aged 18-26) referred to one clinic in Los Angeles, CA. The study site has a wide range of referral sources ranging from self-referral to referrals from the justice system.

Some young adults are referred to treatment by schools in lieu of engaging law enforcement or in lieu of expulsion, with many being self-referred.

Participants will be randomly assigned to receive MBRP or attention control (CTL). Participants will engage in both self-report and task-based ER, IMP, and EF measures pre- and post-intervention. Participants will be followed for 3 months post-intervention to assess effects on alcohol use and behavioral health outcomes, and putative mechanisms of change.

The central hypothesis is that MBRP, compared to CTL, will prompt change in ER, IMP, and EF. Further, it is hypothesized that these changes will be associated with better alcohol use outcomes 3 months post-intervention. The rationale for using a MBI with marginalized youth is that prior research has shown significantly worse self-regulation compared to community youth, and MBRP is specifically designed to aid in regulating emotions, decision making, and attention control. The unique strengths of this proposal are its use of an MBI; focus on a disadvantaged population of diverse racial and ethnic groups; focus on putative targets essential to behavioral health outcomes; and use of multiple neurocognitive tasks addressing important self-regulation components. The study objective is to test following three aims:

Specific Aim 1: Determine feasibility and acceptability of abbreviated MBRP. An adapted MBRP protocol will be beta-tested with 15 transition age youth/young adults. Focus groups will be conducted to evaluate the feasibility and acceptability of an intervention focused on enhancing self-regulation, refine content based on feedback, and addressing issues that might affect the successful completion of pilot testing in Aim 2.

Specific Aim 2: Pilot test MBRP intervention on putative targets by randomly assigning young adults who screen for past-month alcohol use/problems to MBRP or CTL. Determine the effect of the program on secondary outcomes of interest and putative targets for ER, IMP, and EF.

Specific Aim 3: Assess MBRP mechanisms by exploring whether effects of the intervention on our substance use outcomes can be partially explained by changes in target mechanisms: ER, IMP, and EF.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 26 years old at baseline
* English speaking
* Be willing to provide follow-up information
* Report past-month use of alcohol or drugs
* Score 2 or higher on the PC-PTSD scale
* Not currently receiving substance abuse treatment elsewhere
* Not prisoners

Exclusion Criteria:

* Does not speak English
* Receiving treatment from some other facility for substance use.
* Active psychosis symptoms

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Substance Use | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months
  Substance use will be measured using time line follow back approach for 15 different substances. We will ask about days of use and number of times used for each substance in the past month
Change in PTSD symptoms | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months
  Initial screening of PTSD symptoms will be assessed by the Primary Care PTSD Screen for DSM-5 (PC-PTSD-5). We will further assess PTSD symptoms using the PTSD Checklist for DSM-5 (PCL-5). The PCL-5 is a 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual of Mental Disorders (DSM-5) symptoms of PTSD.
Change in Depression | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months
  Depression will be measured with the Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D includes 20 items instructing participants how often they have experienced a variety of symptoms in the past week, ranging from "rarely or none of the time" to "Most or all of the time." The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomology.

SECONDARY OUTCOMES:
Executive Functioning | Baseline, 2 months post-baseline
  Executive functioning will be assessed using the Sustained Attention to Response Task (SART). The SART is a computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target (often the digit 3) presented amongst a background of frequent non-targets (0-2, 4-9).
Emotion Regulation | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months
  Emotion regulation will be assessed using the short-form Difficulties in Emotion Regulation Scale (DERS-18). The DERS-18 asks participants to indicate how often they respond to their emotions in a variety of ways. Response options range on a 5-point scale from 1 (almost never, 0-10%) to 5 (Almost always, 91-100%). To obtain a total score, three items are reverse-scored and responses are summed. Total scores range from 18 to 90. Higher scores indicate greater difficulty regulating emotions.
Impulsivity | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months
  The SUPPS-P measures five components: Lack of premeditation, lack of perseverance, negative urgency, positive urgency, sensation seeking.
Delinquency | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months
  Delinquency will be assessed by self-reported offending.
Stress | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months
  Stress will be assessed using the Perceived Stress Scale (PSS). The PSS is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. The PSS consists of 10 items assessing perceived stress related to a variety of circumstances, with response options for each item existing on a 5-point scale ranging from 0 (never) to 4 (very often). Total PSS scores are obtained by reversing responses to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items (range: 0 to 40). Higher PSS scores reflect higher levels of perceived stress.
Violence Perpetration | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months
  Violence perpetration will be assessed using the Illinois Bullying Scale. Point values are assigned to each response as follows: Never = 0, 1 or 2 times = 1, 3 or 4 times = 2, 5 or 6 times = 3, 7 or more times = 4. Summary scores for each subscale can be obtained by adding the responses for associated items:
  * Bully subscale: Items 1, 2, 8, 9, 14, 15, 16, 17, and 18
  * Victim subscale: Items 4, 5, 6, and 7
  * Fighting subscale: Items 3, 10, 11, 12, and 13
  The Bully subscale score ranges from 0-36; the Victim subscale score ranges from 0-16; and the Fighting subscale score ranges from 0-20). Higher scores reflect higher levels of bullying, victimization, or fighting.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, School of Social Work, Los Angeles, California, United States

REFERENCES:
- [Background] Bechara A, Damasio AR, Damasio H, Anderson SW. Insensitivity to future consequences following damage to human prefrontal cortex. Cognition. 1994 Apr-Jun;50(1-3):7-15. doi: 10.1016/0010-0277(94)90018-3. PMID 8039375
- [Background] Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav. 2014 Sep;39(9):1372-6. doi: 10.1016/j.addbeh.2014.02.013. Epub 2014 Mar 3. PMID 24636739
- [Background] Davis JP, Berry D, Dumas TM, Ritter E, Smith DC, Menard C, Roberts BW. Substance use outcomes for mindfulness based relapse prevention are partially mediated by reductions in stress: Results from a randomized trial. J Subst Abuse Treat. 2018 Aug;91:37-48. doi: 10.1016/j.jsat.2018.05.002. Epub 2018 May 20. PMID 29910013
- [Background] Espelage, D. L., & Holt, M. K. (2001). Bullying and victimization during early adolescence: Peer influences and psychosocial correlates. Journal of Emotional Abuse, 2(2-3), 123-142. https://doi.org/10.1300/J135v02n02_08
- [Background] Hallion LS, Steinman SA, Tolin DF, Diefenbach GJ. Psychometric Properties of the Difficulties in Emotion Regulation Scale (DERS) and Its Short Forms in Adults With Emotional Disorders. Front Psychol. 2018 Apr 19;9:539. doi: 10.3389/fpsyg.2018.00539. eCollection 2018. PMID 29725312
- [Background] Himelstein, S. (2011). Mindfulness-Based Substance Abuse Treatment for Incarcerated Youth: A Mixed Method Pilot Study. International Journal of Transpersonal Studies, 1-10.
- [Background] Himelstein, Sam, Hastings, A., Shapiro, S., & Heery, M. (2012). Mindfulness training for self-regulation and stress with incarcerated youth. Probation Journal, 59(2), 151-165. https://doi.org/10.1177/0264550512438256
- [Background] Himelstein S, Saul S, Garcia-Romeu A, Pinedo D. Mindfulness training as an intervention for substance user incarcerated adolescents: a pilot grounded theory study. Subst Use Misuse. 2014 Apr;49(5):560-70. doi: 10.3109/10826084.2013.852580. PMID 24611851
- [Background] Jackson JD, Balota DA. Mind-wandering in younger and older adults: converging evidence from the Sustained Attention to Response Task and reading for comprehension. Psychol Aging. 2012 Mar;27(1):106-119. doi: 10.1037/a0023933. Epub 2011 Jun 27. PMID 21707183
- [Background] Leonard NR, Jha AP, Casarjian B, Goolsarran M, Garcia C, Cleland CM, Gwadz MV, Massey Z. Mindfulness training improves attentional task performance in incarcerated youth: a group randomized controlled intervention trial. Front Psychol. 2013 Nov 8;4:792. doi: 10.3389/fpsyg.2013.00792. eCollection 2013. PMID 24265621
- [Background] Prins A, Bovin MJ, Smolenski DJ, Marx BP, Kimerling R, Jenkins-Guarnieri MA, Kaloupek DG, Schnurr PP, Kaiser AP, Leyva YE, Tiet QQ. The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5): Development and Evaluation Within a Veteran Primary Care Sample. J Gen Intern Med. 2016 Oct;31(10):1206-11. doi: 10.1007/s11606-016-3703-5. Epub 2016 May 11. PMID 27170304
- [Background] Selner-O'Hagan MB, Kindlon DJ, Buka SL, Raudenbush SW, Earls FJ. Assessing exposure to violence in urban youth. J Child Psychol Psychiatry. 1998 Feb;39(2):215-24. PMID 9669234
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729